CLINICAL TRIAL: NCT02479880
Title: Pharmacoepidemiology Study to Define the Long-term Safety Profile of Tenofovir Disoproxil Fumarate (Tenofovir DF, Viread®) and Describe the Management of Tenofovir DF-associated Renal and Bone Toxicity in Chronic Hepatitis B (CHB)-Infected Adolescents Aged 12 to <18 Years in Europe
Brief Title: Utilization and Efficacy of Tenofovir DF in Adolescents With Chronic Hepatitis B Virus Infection
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: GS-EU-174-1403; 2014-004939-39 (EudraCT Number)
Record Dates: First submitted 2015-06-17; First posted 2015-06-24 (Estimated); Results first posted 2019-05-20 (Actual); Last update posted 2019-05-20 (Actual); Status verified 2019-02

CONDITIONS: Hepatitis B
MeSH Terms: conditions — Hepatitis B | interventions — Tenofovir; Absorptiometry, Photon

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tenofovir DF + increased bone/renal monitoring (Other): Participants will receive tenofovir DF, plus laboratory bone biomarker testing and lumbar spine and whole-body DEXA scans every 24 weeks from baseline to Week 96 (5 scans), and monitoring of renal function at 4 and 12 weeks after baseline and every 12 weeks thereafter. With the exception of an enhanced monitoring protocol for bone and renal outcomes, participants will be managed according to local standards of care.
  Interventions: Drug: Tenofovir DF; Radiation: DEXA Scan
- Tenofovir DF + prespecified bone monitoring (Other): Participants will receive tenofovir DF, plus laboratory bone biomarker testing and lumbar spine and whole-body DEXA scans at baseline, Week 48, and Week 96. With the exception of pre-specified bone monitoring, participants will be managed according to local standards of care.
  Interventions: Drug: Tenofovir DF; Radiation: DEXA Scan

INTERVENTIONS:
Drug: Tenofovir DF — 300 mg tablet administered orally once daily for up to 96 weeks
  Other Names: Viread®
Radiation: DEXA Scan — Dual energy x-ray absorptiometry (DEXA) scans administered at protocol-specified time points

SUMMARY:
The primary objective of this study is to characterize the long term (ie, 96 weeks of follow up) bone safety profile of open-label tenofovir disoproxil fumarate (tenofovir DF) treatment in CHB-infected adolescents. This includes prospectively evaluating and comparing the bone mineral density (BMD) change between CHB-infected adolescents 12 to < 18 years of age treated with tenofovir DF in European treatment centers who are assigned to one of two schedules for renal and bone laboratory monitoring and BMD measurement.

ELIGIBILITY:
Key Inclusion Criteria:

1. 12 to <16 years of age
2. Documented chronic hepatitis B virus (HBV) infection
3. Weight ≥ 35 kg
4. Able to swallow oral tablets
5. Negative pregnancy test for females of childbearing potential
6. Adequate kidney (renal) function
7. Parent or legal guardian of potential study subjects able to provide written informed consent

Key Exclusion Criteria:

1. Previously received tenofovir DF
2. Sexually-active males or females of reproductive potential who are not willing to use an effective method of contraception during the study
3. Females who are pregnant or breastfeeding, or females who wish to become pregnant during the course of the study
4. Known hypersensitivity to tenofovir DF, the metabolites or formulation excipients
5. Any condition (including alcohol or substance abuse) or prior therapy that, in the opinion of the Investigator, would make the subject unsuitable for the study or unable to comply with treatment requirements

Note: Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 12 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2015-07-03 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-04-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (11):
- Cliniques Universitaries Saint- Luc, Departem Pediatrie, Brussels, Belgium
- Hopital Femmes Meres Enfants, Bron, France
- Attikon General Hospital Of Athens, Chaïdári, Greece
- Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy
- Romania (3):
  - Grigore Alexandrescu Childrens Emergency Clinical Hospital, Bucharest
  - Spitatul Clinic de Boli Infectioase Constanta, Constanța
  - Institutul de Gastrenterologie si Hepatologie Iasi, Iași
- Spain (3):
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Sant Joan de Déu, Barcelona
  - Hospital de Meixoeiro, Vigo
- Birmingham Children's Hospital NHS Trust, Birmingham, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in Europe. The first participant was screened on 03 July 2015. The last study visit occurred on 11 April 2018. The study did not achieve targeted enrollment as it was prematurely terminated by the Pharmacovigilance Risk Assessment Committee (PRAC).
Pre-assignment Details: 35 participants were screened.
Groups:
- Tenofovir DF + Increased Bone/Renal Monitoring: One 300 mg tablet given once daily for up to 96 weeks + laboratory bone biomarker testing and lumbar spine and whole-body dual-energy x-ray absorptiometry (DXA) scans every 24 weeks from baseline to Week 96 (5 scans), and monitoring of renal function at 4 and 12 weeks after baseline and every 12 weeks thereafter. With the exception of an enhanced monitoring protocol for bone and renal outcomes, participants were managed according to local standards of care.
- Tenofovir DF + Prespecified Bone Monitoring: One 300 mg tablet given once daily for up to 96 weeks + laboratory bone biomarker testing and lumbar spine and whole-body DXA scans at baseline, Week 48, and Week 96. With the exception of pre-specified bone monitoring, participants were managed according to local standards of care.
Period: Overall Study
Arm/Group | Tenofovir DF + Increased Bone/Renal Monitoring | Tenofovir DF + Prespecified Bone Monitoring
Started | 15 | 15
Completed | 2 | 2
Not Completed | 13 | 13
Not completed — Study Terminated by Sponsor | 13 | 12
Not completed — Pregnancy | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included participants who were randomized into the study and received at least one dose of tenofovir DF.
Groups:
- Tenofovir DF + Increased Bone/Renal Monitoring: One 300 mg tablet given once daily for up to 96 weeks + laboratory bone biomarker testing and lumbar spine and whole-body DXA scans every 24 weeks from baseline to Week 96 (5 scans), and monitoring of renal function at 4 and 12 weeks after baseline and every 12 weeks thereafter. With the exception of an enhanced monitoring protocol for bone and renal outcomes, participants were managed according to local standards of care.
- Total: Total of all reporting groups
Arm/Group | Tenofovir DF + Increased Bone/Renal Monitoring | Tenofovir DF + Prespecified Bone Monitoring | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 14 (1.4) | 14 (1.5) | 14 (1.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 10 | 10 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 12 | 25
  Not Hispanic or Latino | 0 | 1 | 1
  Unknown or Not Reported | 2 | 2 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 2 | 5 | 7
  Black or African American | 5 | 5 | 10
  White | 7 | 4 | 11
  Other | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  Greece | 1 | 1 | 2
  Romania | 4 | 4 | 8
  Belgium | 2 | 2 | 4
  Italy | 1 | 0 | 1
  United Kingdom | 2 | 4 | 6
  France | 2 | 1 | 3
  Spain | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Bone-Related Adverse Events and/or a ≥ 4% Reduction in Bone Mineral Density (BMD) From Baseline to Week 96
Time Frame: Baseline to Week 96
Population: Participants in the Safety Analysis Set (participants who were randomized into the study and received at least one dose of tenofovir DF) with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Tenofovir DF + Increased Bone/Renal Monitoring | Tenofovir DF + Prespecified Bone Monitoring
Number analyzed (Participants) | 15 | 15
percentage of participants | 6.7 | 0

ADVERSE EVENTS:
Time Frame: Up to 96 weeks plus 30 days
Description: Safety Analysis Set included participants who were randomized into the study and received at least one dose of tenofovir DF.
Arm/Group | Tenofovir DF + Increased Bone/Renal Monitoring | Tenofovir DF + Prespecified Bone Monitoring
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 1/15 | 2/15
Other Adverse Events (participants affected / at risk) | 10/15 | 10/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tenofovir DF + Increased Bone/Renal Monitoring (N=15) | Tenofovir DF + Prespecified Bone Monitoring (N=15)
Calcinosis (General disorders) | 1 | 0
Malaise (General disorders) | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tenofovir DF + Increased Bone/Renal Monitoring (N=15) | Tenofovir DF + Prespecified Bone Monitoring (N=15)
Abdominal pain (Gastrointestinal disorders) | 1 | 2
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Anal fissure (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Dyschezia (Gastrointestinal disorders) | 1 | 0
Food poisoning (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 0
Fatigue (General disorders) | 0 | 1
Pyrexia (General disorders) | 2 | 0
Hypersensitivity (Immune system disorders) | 1 | 0
Ear infection (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 2 | 0
Otitis media (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 1
Viral infection (Infections and infestations) | 0 | 1
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 1
Bone density decreased (Investigations) | 0 | 2
Vitamin D decreased (Investigations) | 2 | 2
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle contracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 2
Somnolence (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 1 | 0
Dyspareunia (Reproductive system and breast disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (3):
  • Study Protocol: Original (2014-11-03): https://cdn.clinicaltrials.gov/large-docs/80/NCT02479880/Prot_000.pdf
  • Study Protocol: Amendment 2 (2015-03-10): https://cdn.clinicaltrials.gov/large-docs/80/NCT02479880/Prot_001.pdf
  • Statistical Analysis Plan (2018-05-13): https://cdn.clinicaltrials.gov/large-docs/80/NCT02479880/SAP_002.pdf